CLINICAL TRIAL: NCT02986581
Title: Prospective Cohort Study of Rapid Response Team
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SAFER_20161101
Record Dates: First submitted 2016-11-04; First posted 2016-12-08 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Hospital Medical Emergency Team; Medicine, Emergency; Hospital Rapid Response Team
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect data of rapid response team activated patients prospectively

DETAILED DESCRIPTION:
acutely deteriorating patients including sudden cardiac arrest in general ward who are monitored and intervened by rapid response team

ELIGIBILITY:
Inclusion Criteria:

- Patients admitted to general ward in Seoul National University Bundang Hospital and monitored by in-hospital rapid response system.

Exclusion Criteria:

* patients admitted to pediatric wards
* patients in emergency room, intensive care unit, and operating room

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to general ward in Seoul National University Bundang Hospital and monitored by in-hospital rapid response system.
Sampling Method: Non-Probability Sample
Enrollment: 79800 (Estimated)
Dates: Start 2016-11; Primary Completion 2022-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
mortality or ICU admission of rapid response team activated patient | an average of 1 year
incidence of preventable cardiac arrest | an average of 1 year

SECONDARY OUTCOMES:
Frequency of triggerring criteria(1) for activation of rapid response team | an average of 1 year
  SBP <90mmHg(mABP 60mmHg) +- clinically correlated symptom or sign
Frequency of triggerring criteria(2) for activation of rapid response team | an average of 1 year
  HR: <50/min or >140/min or symptomatic arrythmia
Frequency of triggerring criteria(3) for activation of rapid response team | an average of 1 year
  RR: <10/min or >30/min or stridor(sign of airway obstruction) or accessary muscle use
Frequency of triggerring criteria(4) for activation of rapid response team | an average of 1 year
  Oxygenation: SaO2 <90% in room air or FM 8L/min
Frequency of triggerring criteria(5) for activation of rapid response team | an average of 1 year
  Metabolic acidosis: Lactic acid<2.5 , TCO2 <15
Frequency of triggerring criteria(6) for activation of rapid response team | an average of 1 year
  ABGA abnormality : PaCO2>50 or pH<7.3 or PaO2<60
Frequency of triggerring criteria(7) for activation of rapid response team | an average of 1 year
  ABGA abnormality : PaCO2>50 or pH<7.3 or PaO2<60
Frequency of triggerring criteria(8) for activation of rapid response team | an average of 1 year
  Any serious concern about overall deterioration detected by doctor, nurse and caregiver at bedside

CONTACTS AND LOCATIONS:
Overall Officials: Yeon Joo Lee, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea